CLINICAL TRIAL: NCT05915650
Title: Application of PNE in Postoperative Pain Management of Patients With Primary Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Yongmei Zhang, Study Director, Zunyi Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KLLY-2020-147
Record Dates: First submitted 2023-06-01; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education Group (Experimental)
  Interventions: Behavioral: Pain Neuroscience Education
- Routine Education Group (Experimental)
  Interventions: Behavioral: Routine Education

INTERVENTIONS:
Behavioral: Pain Neuroscience Education — Carry out pain neuroscience education intervention for TKA patients
  Arms: Pain Neuroscience Education Group
Behavioral: Routine Education — Carry out routine education intervention for TKA patients
  Arms: Routine Education Group

SUMMARY:
This study intends to carry out pain neuroscience education intervention for TKA patients to clarify the effect of this method on the degree of postoperative pain, the incidence of pain catastrophizing, kinesiophobia, and knee joint function rehabilitation in TKA patients, so as to provide a basis for clinical nursing of such patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as KOA according to the criteria and undergoing unilateral total knee arthroplasty for the first time;
2. The subjects included in this study were men or women aged 45-74 years;
3. Clear self-cognition, can browse the text by themselves or can answer questions correctly;
4. Those who voluntarily participated in the study and signed an informed consent form after understanding the relevant information of the study;
5. Without serious physical diseases such as heart, liver or kidney;
6. No history of mental illness or drug dependence.

Exclusion Criteria:

1. Combined with severe trauma in other parts;
2. Accompanied by serious damage to other organs, such as heart and cerebrovascular diseases, lung and kidney diseases;
3. Patients with knee tumor and severe knee deformity who could not complete the rehabilitation;
4. With neurological diseases that limit physical activity;
5. Participating in other investigators during the same period.

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale pain score, (VAS) | 3 months after discharge
  Status of pain

CONTACTS AND LOCATIONS:
Locations (1):
- Yongmei Zhang, Zunyi, Guizhou, China